CLINICAL TRIAL: NCT01645215
Title: Phase I Study of Safety and Pharmacokinetics of Fruquintinib(HMPL-013) in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Fruquintinib(HMPL-013) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-013-00CH1
Record Dates: First submitted 2012-03-15; First posted 2012-07-20 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2013-09

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fruquintinib capsule (Experimental): cohort 1: fruquintinb continuous oral dosing (1mg once a day) cohort 2: fruquintinb continuous oral dosing (2mg once a day) cohort 3: fruquintinb continuous oral dosing (4mg once a day) cohort 4: fruquintinb continuous oral dosing (6mg once a day) cohort 5: fruquintinb continuous oral dosing (5mg once a day) cohort 6: fruquintinb oral dosing, 3 weeks on/1 week off (5mg once a day) cohort 7: fruquintinb oral dosing, 3 weeks on/1 week off (6mg once a day)
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib is a capsule in the form of 0.25mg , 1mg and 5mg, oral, once a day.
  Other Names: HMPL-013

SUMMARY:
Fruquintinib (HMPL-013) is a novel oral small molecule that selectively inhibits vascular endothelial growth factor receptors (VEGFR) 1, 2, and 3 and has demonstrated potent inhibitory effects on multiple human tumor xenografts. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics , safety and preliminary anti-tumor activity of HMPL-013 at single doses and multiple doses .

DETAILED DESCRIPTION:
This will be an open-label, phase I study. This study will evaluate the safety and pharmacokinetics of HMPL-013 after a single administration followed by a 28-Day continuous course of therapy; evaluate the safety and preliminary efficacy in an open-label administration of at the MTD. All subjects of this study will be permitted to continue therapy with only safety monitoring and bimonthly assessments for progression, if the product is well tolerated and the subject has stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histological or cytological confirmed solid malignant tumor
* ECOG performance status of 0-1
* Standard regimen failed or no standard regimen available
* Life expectancy of more than 12 weeks
* LVEF ≥ 50%
* Duration from the last therapy is more than 4 weeks for operation or radiotherapy; more than 4 weeks for prior systemic treatment
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 × 109/L, neutrophil > 1.5 × 109/L, hemoglobin > 90g/dl ,serum creatinine within upper limit of normal(ULN), total bilirubin and serum transaminase within upper limit of normal(ULN), and PT, APTT, TT, Fbg normal
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure

Exclusion Criteria:

* Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Evidence of uncontrolled CNS metastasis
* Intercurrence with one of the following: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial
* Previous treatment with VEGF/VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Proteinuria ≥ 2+
* Uncontrolled hemorrhage in GI
* Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Within 6 months before the first treatment occurs acute myocardial infarction, acute coronary syndrome or CABG
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety in the first 28-Days of Therapy | 28-Days after Permanent Discontinuation of HMPL-013
  The primary endpoint is evaluation of safety during the first 28-day cycle of therapy following the initiation of multiple dosing of HMPL-013. The safety variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology , and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate.

SECONDARY OUTCOMES:
Objective Response Rate （ORR) | every 8 weeks until end of treatment
  Anti-tumoral efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors (RECIST v 1.0) at baseline (Day -14 to -1) and at the end of two 28-Day cycles of therapy . For patients that continue on repeat 28-Day cycles after the primary evaluation period, progression will be assessed after each two 28-Day cycles of therapy.
Pharmacokinetic Assessments for AUC, Cmax and Tmax | Day 1-3 Single Dose and Day 1-28 Steady State
  In the study of single-dose, full PK profiles of HMPL-013 will be obtained following administration of a single oral dose of HMPL-013 on Day 1 to Day 3. At multiple-dose, PK sampling will include a pre-dose and at the 1,4,8,12 hour time points on days 1,14,28 of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2, 3, 7, 15 and 29 of the first 28-Day cycle of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China